CLINICAL TRIAL: NCT04730830
Title: Survenue Des Infections d'Emergence après la Pose d'un catHéter de Dialyse péritonéaLE
Brief Title: Occurrence of Emerging Infections After Placement of a Peritoneal Dialysis CatHeter
Acronym: SINEPHILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/504
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: End Stage Renal Disease on Dialysis; Peritoneal Dialysis
Keywords: Renal disease; Peritoneal dialysis; Emergence infections
MeSH Terms: conditions — Kidney Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Observational study with questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only experimental arm (Experimental): Only experimental arm. Patients filling out questionnaires.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients completing emergence assessment questionnaires at the time of the first dressing placement, as well as at the scheduled weekly placement. As part of a planned repair, the emergence will be assessed at most once a week, preferably at the beginning of the week by the patient. In any other case of dressing change, an emergence assessment will be requested.

SUMMARY:
Peritoneal dialysis, which appeared at the end of the 1970s, quickly proved its worth both in terms of its effectiveness and of its ease of compliance, which guarantees an improved quality of life. To date there are different modes of application of this technique: Continuous Ambulatory Peritoneal Dialysis, and Automated Peritoneal Dialysis. Whatever the technique used, the placement of a dressing covering the exit site of the catheter is necessary just after the placement of the PD catheter and this so that the site of emergence is kept dry until healing (in general 2 to 4 weeks). Once the emergence site has healed, the technique can be started. Discharge site infections are a major predisposing factor for the development of peritonitis. Numerous studies in different parts of the world have shown that the rates of PD-related infections have steadily declined over the past 10 to 20 years. Several recommendations for the prevention and treatment of emergence site infections have been published by the International Peritoneal Dialysis Society. Several studies nonetheless call into question the recommendations by showing that catheter infection is not linked to the number of risk factors present at the time of catheter insertion, nor to the prescription of antibiotic prophylaxis, nor to the the experience of the caregiver, the antiseptic used or the early dressing change. In addition, only antibiotic prophylaxis at catheter placement is strongly recommended. Regarding the other measures, their relevance is not always demonstrated and their application varies considerably from one center to another. In addition, many authors have sought to establish a definition of catheter infections in order to allow an optimal assessment of their frequency. However, these definitions are not universal and have certain limitations. The objective of this work is on the one hand to better characterize the incidence of infections at the site of emergence in peritoneal dialysis, and on the other hand, in the absence of a definition established according to the recommendations, to use the score de Schaeffer, is in particular the value of this score which would make it possible to define more precisely the presence of an infection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 inclusive
* Signature of informed consent
* Affiliation to a French social security scheme
* Patient with end stage renal disease starting renal replacement therapy by peritoneal dialysis in one of the participating centers

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Pregnant woman
* Subject being in the period of exclusion from another study or provided for by the "national file of volunteers".
* Patient without health insurance
* Inability to understand the reasons for the study; psychiatric disorder judged by the investigator to be incompatible with inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Risk of infections on emergence site | 24 months
  The risk of infections on emergence site of placing a peritoneal dialysis catheter. The infection of the site of emergence is defined by the practitioner as a minimum according to the recommendations: "the presence of a purulent discharge, with or without erythema of the skin at the catheter-epidermal interface" and inducing treatment with an antibiotic .

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de néphrologie, CHU de Besançon, Besançon
  - Besancon University Hospital, Besançon